CLINICAL TRIAL: NCT04246736
Title: Bädda för Kvalitet: Proaktiva Strategier för återhämtning i främjandet av hälsa Och Arbetsprestation.
Brief Title: A Proactive Intervention Promoting Strategies for Sleep and Recovery in Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: AFA Insurance (Industry)
Responsible Party: Principal Investigator, Anna Dahlgren, Project manager, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AFA:150024
Record Dates: First submitted 2019-12-17; First posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Sleep; Occupational Stress; Fatigue; Behavior, Health; Burnout; Sleepiness; Shift-Work Related Sleep Disturbance; Cognitive Symptom; Insomnia
Keywords: sleep; fatigue; stress; recovery; occupational; shiftwork; strategies; work performance; burnout; sleepiness; newly graduated nurses
MeSH Terms: conditions — Occupational Stress; Fatigue; Health Behavior; Burnout, Psychological; Sleepiness; Neurobehavioral Manifestations; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Participants were randomised into intervention group and control group. The intervention group received the intervention and were followed-up until 6 months after the intervention. After that, the control group received the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group received a "Recovery programme" including three group sessions.
  Interventions: Behavioral: Bädda för Kvalitet
- Control group (No Intervention): The control group was on a waiting list to receive the intervention after the last follow-up measure (six months after the intervention group's last group session).

INTERVENTIONS:
Behavioral: Bädda för Kvalitet — A group-administered preventive programme focusing on beneficial strategies for sleep and recuperation, in relation to work related stress and shift work. The intervention was based on knowledge from previous research on sleep, stress and work hours, as well as on cognitive behavioural therapy (CBT) techniques for sleep and stress management, modified for shift workers. Participants were encouraged to discuss and reflect on personal habits related to sleep and recovery. As homework between sessions, the participants were encouraged to try possibly beneficial strategies for sleep and recuperation. All participants got written material covering the content of the session, during each sessions. In addition, an adapted version of a biomathematical model ("ArturNurse") was used to give participants an estimation of expected sleep lengths and fatigue levels together with tips of possible strategies to optimise sleep in relation to different shifts.
  Arms: Intervention group

SUMMARY:
Considering the known challenges facing newly graduated nurses, there are possibilities to implement preventive actions. The aim of the current study was to evaluate the effects of a preventive intervention among newly graduated nurses, supporting proactive strategies for sleep and recuperation in relation to work related stress and shift work.

DETAILED DESCRIPTION:
Approximately 20% of all Swedish nurses experiences very high levels of burnout symptoms at some point during the first years of practice. Many factors are likely to be involved, and when developing methods to facilitate the nurse's transition from education into working life, a variety of stressors at both the organisational and individual level have to be considered. Previously, incomplete recovery has been suggested to mediate the relation between stressful working conditions and health impairment. For many, starting working as a nurse also means an introduction to shiftwork, which inevitably affects opportunities for sleep and recuperation due to interference with the circadian and homeostatic regulation of sleep. Given the vital role of sleep and recovery in the relationship between stress and development of impaired health, effective strategies for sleep and recuperation are hypothesised to be crucial in preventing the development of stress-related symptoms among nurses. In addition, lack of sleep and recuperation results in fatigue, which is a major safety hazard threatening patient safety. The aim of the current study was to evaluate a preventive intervention for new nurses, supporting strategies for sleep and recuperation in relation to work related stress and shift work.

Recruitment Newly graduated nurses were recruited at five Swedish hospitals. The recruitment was done via the introduction programmes, except from at one of the hospitals (which did not have such a programme) where the nurses instead were recruited via the different clinics. In total the intervention was implemented in eight different cohorts during 2017 and 2018. Approximately 462 newly graduated nurses were invited to participate in the study and 207 joined and answered the baseline questionnaire (45%).

Design The participants were randomly assigned to intervention and control groups. The participants were followed with questionnaires Participants were followed with either questionnaires or questionnaires + intesive measures using diary, actigraphy and cognitive tests. Questionnaires were filled in before the intervention (baseline), one month after the intervention (post), and at six months after the intervention (follow-up). The intensive measure was conducted at baseline and post intervention.

The participants also got a short questionnaire to fill out at the start of session two and three, and two weeks after session three, in which they filled out which strategies they had used during the last couple of weeks. After the last session, participants were asked to evaluate the intervention using a short questionnaire.

The intervention The intervention was a preventive programme focusing on beneficial strategies for sleep and recuperation in relation to work stress and shift work. The programme included three 2.5 hours-group sessions every second week. The sessions were taking place at work during working hours. The intervention was based on knowledge from research on sleep, stress and work hours, as well as on cognitive behavioural therapy (CBT) techniques for sleep and stress management modified for shift workers. The regulation of sleep and wakefulness was explained by the three factors: 1) circadian rhythm, 2) homeostatic process, and 3) stress, referred to as the sleep formula. How these factors interacts with irregular work hours was explained. Participants were encouraged to reflect on their daily habits related to sleep and recovery. Also, a CBT-model for analysing behaviours in stressful work situations were used in order to encourage participants to reflect on their usual behaviours and possible alternatives. As homework between sessions, the participants were encouraged to try possibly beneficial strategies for sleep and recuperation. The participants got written material, after every session, covering the content of the session. In addition, the participants got access to an adapted version of the biomathematical model (ArturNurse) to give participants an estimation of expected sleep lengths and fatigue levels together with tips of possible strategies to optimise sleep in relation to different shifts.

ELIGIBILITY:
Inclusion Criteria:

* Newly graduated nurse in the first year of employment

No Exclusion Criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2018-12-13 (Actual)

PRIMARY OUTCOMES:
Change in insomnia symptoms (subjective measure) | In order to detect change measures were made at baseline, 4 weeks after the intervention and 6 months after the intervention.
  Insomnia Severity Index (ISI) which consists of 7 questions related to sleep e.g. "How satisfied are you with your current sleep pattern?" (0 = very satisfied, 4 = very dissatisfied). The total score is summarised with a minimum score 0, maximum score 28. Higher scores indicate more sleep problems.
Change in sleep quality (subjective measure) | In order to detect change measures were made at baseline, 4 weeks after the intervention and 6 months after the intervention.
  Karolinska Sleep Questionnaire (KSQ) from which a sleep quality index was formed based on four questions e.g. "Have you had problems falling asleep the past month"? etc : Minimum score 1, maximum score 6. Lower scores indicate worse sleep quality.
Change in Dysfunctional beliefs and attitudes about sleep (subjective measure) | In order to detect change measures were made at baseline, 4 weeks after the intervention and 6 months after the intervention.
  Dysfunctional Beliefs and Attitudes about Sleep (DBAS) consists of 10 statements regarding beliefs and attitudes to sleep e.g. "I am concerned that chronic insomnia may have serious consequences on my physical health"; "When I have trouble sleeping, I should stay in bed and try harder" (strongly agree - strongly disagree): Minimum score 0, maximum score 10. Higher scores indicate more dysfunctional sleep-related cognitions.
Change in sleep (subjective measure) | In order to detect change measures were made at baseline to 4 weeks after the intervention. Measured seven days at baseline and seven days at follow up.
  Karolinska Sleep Diary (KSD). KSD includes bedtime; time of awakening; sleep latency (the time it takes to fall asleep); feelings of worry and stress at bedtime (1 very worried/aroused - 5 very calm/relaxed); and the following questions: Did you have difficulties falling asleep? (1 = very; 5 = not at all) How did you sleep? (1 = very badly; 5 = very good); Did you have a restless sleep? (1 = very much so; 5 = not at all); Did you wake up very early without being able to fall asleep? (1 = much too early; 5 = no). These four latter questions constitutes a sleep quality index, minimum score 1, maximum score 5: Lower scores indicate worse sleep quality.
Change in satisfaction with sleep | In order to detect change measures were made at baseline, 4 weeks after the intervention and 6 months after the intervention.
  Self-rated sufficient sleep (5=very insufficient 1=fully sufficient)
Change in subjective sleep quality | In order to detect change measures were made at baseline, 4 weeks after the intervention and 6 months after the intervention.
  Self-rated general sleep quality (1=very good 5=very bad).
Change in sleep (objective measures) | In order to detect change measures were made at baseline and at 4 weeks after the intervention. Measured seven days at baseline and seven days at follow up.
  Actigraphy (wrist-watch). Measuring of movements during sleep through a sensitive accelerometer in the wrist-watch. The value, which is described as the amount of movements per minute, is saved in the memory of the actigraph. Preprogrammed algorithms make it possible to classify if the participant has slept or not. Measured seven nights at baseline and seven nights at follow up. Example of measures:
  Actual sleep time: The total time spent in sleep according to the epoch-by-epoch wake/sleep categorisation.
  Actual sleep %: Actual sleep time expressed as a percentage of the assumed sleep time.
  Actual wake time: The total time spent in wake according to the epoch-by-epoch wake/sleep categorisation.
  Wake bouts: The number of contiguous sections categorised as wake in the epoch-by- epoch wake/sleep categorisation.
  Sleep fragmentation: The sum of the "Mobile time (%)" and the "Immobile bouts <=1min (%)". This is an indication of the degree of fragmentation.
Change in work home interference (subjective measures) | In order to detect change measures were made at baseline, 4 weeks after the intervention and 6 months after the intervention.
  Work-Home Interference (WHI) measured with four items: "I come home from work too tired to do things I would like to do."; "My job makes it difficult to maintain the kind of personal life I would like."; "I often neglect my personal needs because of the demands of my work."; "My personal life suffers because of my work." Rated on a 5-graded scale ranging from 1=not at all to 5=almost always.
Change in fatigue and recuperation (subjective measures) | In order to detect change measures were made at baseline, 4 weeks after the intervention and 6 months after the intervention.
  Single items (self-ratings): Frequency of recovery behaviours (e.g. micro breaks (1 = every shift, 5 = Never); routine for winding down before bedtime (1 = never, 5 = Always); Satisfaction regarding rest and recuperation during spare time (1 = fully sufficient, 5 = no, far from sufficient); Use of strategies for optimizing sleep and recuperation (1 = never, 5= always); General satisfaction with spare time (1 = very good, 5 = very bad); Use of free time before evening shifts (1 = never, 5 = always); Frequency of breaks during work shifts (1 = every shift, 5= never).
Change in diurnal levels of sleepiness (subjective measures) | In order to detect change measures were made at baseline and 4 weeks after the intervention.
  Karolinska Sleepiness Scale (KSS): A nine-graded scale with values ranging from 1=very alert to 9=very sleepy, fighting sleep. Measured every third hour during wake time seven days at baseline and seven days at follow up.
Change in symptoms of sleepiness and fatigue (subjective measures) | In order to detect change measures were made at baseline to 4 weeks after the intervention.
  Single items measuring symptoms of fatigue e.g. "sustained fatigue", "unfocused" and "engaged", on a five-graded scale ranging from 1=not at all, and 5=very much. Measured seven days at baseline and seven days at follow up.
Change in burnout (subjective measure) | In order to detect change measures were made at baseline, 4 weeks after the intervention and 6 months after the intervention.
  Shirom-Melamed Burnout Questionnaire (SMBQ): Minimum score 1, maximum score 7. Higher scores indicate more burnout.
Change in perceived stress (subjective measure) | In order to detect change measures were made at baseline, 4 weeks after the intervention and 6 months after the intervention.
  Perceived Stress Scale (PSS-10) which consists of 10 statements e.g.. "In the last month, how often have you felt nervous and "stressed"; "In the last month, how often have you found that you could not cope with all the things that you had to do"? etc: Answers on 0 = never, 4 = very often. These are summarised. Minimum score 0, maximum score 40. Higher scores indicate more stress.
Change in stress and energy (subjective measures) | In order to detect change measures were made at baseline and 4 weeks after the intervention.
  Stress-Energy rating questionnaire: Minimum score 0, maximum score 5. Higher scores indicate more stress and more energy.
Change in stress symptoms (subjective measures) | In order to detect change measures were made at baseline and 4 weeks after the intervention.
  Self-ratings of stress symptoms/absence of stress symptoms (single items): "Tense"; "Irritated"; "Exhausted"; "Hard to disconnect from thoughts of work during spare time"; "Emotional burden"; "Relaxed/calm" on a scale ranging from 1=not at all, and 5=very much. Measured every day during seven days at baseline and seven days at follow up.
Change in diurnal levels of stress (subjective measures) | In order to detect change measures were made at baseline and 4 weeks after the intervention.
  Self-rated stress scale for repeated measurement, measured one a nine-graded scale with values ranging from 1=very low stress to 9=very high stress. Measured every third hour during wake time seven days at baseline and seven days at follow up.
Change in stress (objective measures) | In order to detect change measures were made at baseline and 4 weeks after the intervention.
  Hair cortisol based on 2 cm segments (pg/mg)
Change in somatic symptoms | In order to detect change measures were made at baseline, 4 weeks after the intervention and 6 months after the intervention.
  Somatic Symptoms Scale-8 (SSS-8): Minimum score 0, maximum score 32. Higher scores indicate higher somatic symptom burden.
Change in health | In order to detect change measures were made at baseline, 4 weeks after the intervention and 6 months after the intervention.
  Single items: Self-rated health on a scale ranging from 1=very good to 7=very bad. Self-rated use of medical drugs the past three months (frequency as 1 = never, 5 = always), coffee consumption during a work day (1 = none, 5 = 7 cups or more); how often do you do 30 minutes of physical exercise (1 = never, 5 = 3 times of more/week).
Change in psychological health | In order to detect change measures were made at baseline, 4 weeks after the intervention and 6 months after the intervention.
  Single items (self-ratings): How often have you during the past 7 days felt "depressed"; "stated"; "sad"; "worried"; "nervous"; "unsure" on a scale ranging from 0=not at all to 5=very much.
Change in self rated health | In order to detect change measures were made at baseline and 4 weeks after the intervention.
  Self-rated health on a scale ranging from 1=very good to 7=very bad. Measured daily during seven days at baseline and seven days at follow-up.
Change in performance and cognitive symptoms (subjective measures) | In order to detect change measures were made at baseline, 4 weeks after the intervention and 6 months after the intervention.
  Ratings (single items): Self-rated work performance through the following items: During the past month how often have you during you work .... "in risk of mistakes"; "found it hard to make decisions"; "been present during interaction with others"; "had to make corrections or double-check work tasks" (1 = never, 5 = Always). Sub-indices from SMBQ (described above) will also be used as measures of cognitive symptoms.
Change in performance and cognitive symptoms (subjective measures) | In order to detect change measures were made at baseline and 4 weeks after the intervention. Measured seven days at baseline and seven days at follow up.
  Self-ratings (single items) of how well the participant managed to (at work) make decisions; keep things in their head; keep track of the overall picture; perform tasks in a safe way; being present during interaction with others. Rated on a 5-graded scale ranging from 1=very well to 5=very badly.
Change in performance, arithmetic ability (objective measures) | In order to detect change tests were made at baseline (one day, during and after work) and 4 weeks after the intervention (one day, during and after work).
  Cognitive tests measuring executive functioning, performed on the participant's mobile phone. In the arithmetic ability task, the participant is presented with simple arithmetical addition questions and required to calculate the answer and type it into the phone. New questions are presented until the time is running out (duration 2 minutes). Performance is measured in terms of total score (correct responses during 2 minutes) and the speed of correct responses (in ms).
Change in performance, episodic memory (objective measures) | In order to detect change tests were made at baseline (one day, during and after work) and 4 weeks after the intervention (one day, during and after work).
  Cognitive tests measuring executive functioning, performed on the participant's mobile phone. In the episodic memory task, participants are presented with a list of 12 words for 12 seconds, which they are asked to remember. A fixation cross then appears for 5 seconds. Following this, participants are shown a list of 24 words, which contains the original 12 words, and an additional 12 dummy words, and are asked whether each word was previously shown (yes/no). The task is performed twice. Performance is assessed as percentage correct.

SECONDARY OUTCOMES:
Changes in work measures | Baseline, 4 weeks after the intervention and 6 months after the intervention.
  Single items (self-ratings): Satisfaction with work; Work environment ratings (e.g. tempo, emotional demands, control over work tasks, support, engagement, frequency of tasks in conflict with personal values, quality of cooperation with coworkers); Self-rated patient safety at workplace; Work time control (WTC) where the respondents rate on a five graded scale (1=very little to 5=very much) how much they are able to influence the following aspects of their working times: length of a work shift, the starting and ending times of a work shift, the taking of breaks during the work shift, the scheduling of work shifts, the scheduling of vacations and days off, and the handling of private matters during the workday
Changes in working hours | Baseline, 4 weeks after the intervention and 6 months after the intervention.
  Single items (self-ratings):
  Frequency (per month) of overtime work, night shifts and quick returns (less than 11 hours between shifts). Self-rated experiences of problems regarding these different type of shifts/shift combinations (yes/no), type of shift schedule, satisfaction with working hours (1 = very bad, 5 = very good).

CONTACTS AND LOCATIONS:
Locations (7):
- Sweden (7):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Karolinska Universitetssjukhuset, Huddinge
  - Universitetssjukhuset, Linköping
  - Lasarettet Ljungby, Ljungby
  - Vrinnevisjukhuset, Norrköping
  - Karolinska Universitetssjukhuset, Solna
  - Centrallasarettet, Vaxjo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dahlgren A, Tucker P, Epstein M, Gustavsson P, Soderstrom M. Randomised control trial of a proactive intervention supporting recovery in relation to stress and irregular work hours: effects on sleep, burn-out, fatigue and somatic symptoms. Occup Environ Med. 2022 Jul;79(7):460-468. doi: 10.1136/oemed-2021-107789. Epub 2022 Jan 24. PMID 35074887